CLINICAL TRIAL: NCT04077996
Title: Randomized Multicentric Clinical Trial, Efficcacy of the Treatment Application on Peritonitis in Automated Peritoneal Dialysis (APD); Comparision Between APD Versus Ambulatory Dialysis.
Brief Title: Treatment of Peritonitis in Automated Peritoneal Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Colima (Other)
Collaborators: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, J JESUS VENEGAS, D. Sc., Master Degree, Universidad de Colima
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01APDPERITONITIS
Record Dates: First submitted 2019-09-01; First posted 2019-09-04 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Secondary Peritonitis
Keywords: PERITONITIS; AUTOMATED PERITONEAL DIALYSIS; TREATMENT OF PERITONITIS
MeSH Terms: conditions — Peritonitis | interventions — Peritoneal Dialysis, Continuous Ambulatory

STUDY DESIGN:
Intervention Model Description: Patients will be randomly through table of random numbers, and divided to form two treatment groups with 32 patients per group. One of which will be a APD and the other a CAPD + APD. The initial antibiotic scheme will be applied to both groups continuously based on: ceftazidime (1500-2000mg/day) and vancomycin (20mg/kg every 3 days) according to current management guidelines;
Who Masked: Outcomes Assessor
Masking Description: the outcomes assessor will mask to do statistical analisis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peritonitis treatment with one exchange in CAPD (Active Comparator): This group will receive peritonitis treatment with one exchange on Continuous Ambulatory Peritoneal Dialysis per day. The initial antibiotic scheme will be with ceftazidime (1500mg/day) and vancomycin (20mg/kg every 3 days) according to current management guidelines; adjusting the management according to the result of the culture, completing the antibiotic scheme for 14 to 21 days.
  Interventions: Device: Peritonitis treatment with one exchange in CAPD
- Peritonitis treatment placed in APD (Experimental): This group will receive peritonitis treatment placed in Automated Peritoneal Dialysis. The initial antibiotic scheme will be with ceftazidime (1500mg/day) and vancomycin (20mg/kg every 3 days); adjusting the management according to the result of the culture, completing the antibiotic scheme for 14 to 21 days.
  Interventions: Device: Peritonitis treatment placed in APD

INTERVENTIONS:
Device: Peritonitis treatment placed in APD — Antibiotic treatment of peritontiis placed in bags of Automated peritoneal dialysis.
  Arms: Peritonitis treatment placed in APD
Device: Peritonitis treatment with one exchange in CAPD — Antibiotic treatment of peritontiis placed in one bag of Continuos ambulatory peritoneal dialysis per 6 hours each day.
  Arms: Peritonitis treatment with one exchange in CAPD

SUMMARY:
The main infectious complication of peritoneal dialysis (PD) is bacterial peritonitis, which increases morbidity, mortality and conversion to hemodialysis.

In Mexico, 485 patients per million people undergo PD. The Mexican Institute of Social Security (IMSS) reported 55,101 patients with kidney failure, 59% on PD. Automated PD (APD) has contributed by reducing peritonitis. The treatment of peritonitis in APD is carried out by changing to continuous ambulatory peritoneal dialysis (CAPD) or by adding a CAPD/day replacement, increasing costs and delaying treatment. OBJECTIVE: To compare the efficacy of peritonitis antibiotic treatment applied in a DPA bag versus applied in a CAPD/day replacement plus APD in IMSS beneficiaries. MATERIAL AND METHODS: A non-inferiority, multicenter clinical trial was carried out with patients> 18 years of age in APD with peritonitis. Group 1 (g1) receives antibiotics in DPA bags, group 2 (g2) receives antibiotics in a CAPD / day exchange plus APD. The antibiotics applied were ceftazidime 1500 mg / day 14 days and vancomycin 20 mg / kg every 3 days, 5 doses adjusted according to culture, followed by cytology every 48 hours until clinical resolution. Considering resolved peritonitis when symptoms disappeared and white blood cells <100 cells / mm3 were obtained in cytology. The Research and Ethics Committee approved the study. Relative risk (RR), relative risk reduction (RRR) were calculated. The Chi squared test, Student's t test, non-inferiority analysis was calculated considering p <0.05 significant, SPSS 24 and Epi Info were used.

DETAILED DESCRIPTION:
GENERAL DESCRIPTION OF THE STUDY.

PROCEDURES:

Patients with peritonitis (clinical, cytological sample with leukocytes >100/μL, and >50% Polymorphonuclear, taken from a dialysis exchange with 2 to 4 h of stay in the cavity, gram positive or positive culture of dialysis fluid) in Automated peritoneal dialysis of the general hospitals of the Mexican Institute zone Social Security No. 1, 10 and subzone 4 in the state of Colima. Two groups each of 32 patients were forming. Both created treatment groups received antibiotic management based on a double antibiotic scheme with Vancomycin and Ceftazidime via intraperitoneal (IP), the difference was for the treatment group (group 1) the application of the antibiotic through the 6L bags in APD through the cycler machine versus for the control group (group 2) the addition of a manual exchange (CAPD) of 6 hours of stay in extra cavity during the day for the application of the antibiotic plus the

Usual APD at night, the management of peritonitis in each group was established according to the following way:

* Group 1: IP antibiotic treatment applied inside DPA bags. Applied Vancomycin-based antibiotic 20 mg/kg every 72 hours (3 days) applied to bags of DPA (50% in each bag of the total dose) in night exchange every 3 days completing 5 doses, and Ceftazidime 1500mg applied in bags of DPA (50% in each bag of the total dose) each day for 14 days.
* Group 2: IP antibiotic treatment applied to one manual exchange (CAPD) per day, with a stay of 6 hours plus usual DPA programmed at night. The dose administered was Vancomycin 20 mg/kg every 72 hours (3 days) completing 5 dose, and Ceftazidime 1500 mg/day in a manual exchange with a stay of 6 hours for 14 days plus the usual prescribed DPA at night.
* Both groups received training and reviewed the correct application of the antibiotic by the nursing staff of the peritoneal dialysis service during hospitalization or at appointments in the peritoneal dialysis program.
* The researchers and staff of the dialysis program maintained a follow-up of the cases during their stay in hospital, through home visits, phone call and check-up medical appointment.

Patients and relatives were informed in detail about the research project companions mentioning the objectives, risks and benefits of this, their Authorization for inclusion in the study by signing an endorsed informed consent by the national ethics and research committee of the IMSS. Through direct interview and review of the medical record, general and demographic data, data on associated pathologies, comorbidities, time in management with peritoneal dialysis, time of APD management, number of peritoneal catheters placed, APD prescription, diuresis residual, dose of erythropoietin, onset of the clinical picture of peritonitis, as well as the characteristics of the initial frame, time elapsed from the beginning of the frame to the performance of cytology. Possible triggering causes of the symptoms of peritonitis, the peritoneal dialysis technique was verified, other probable sites of infection and close contact was maintained with the medical team in charge of managing the cases hospitalized. After the diagnosis or suspicion of the case of peritonitis, a culture of fluid was taken from dialysis (LD) without antibiotics, and was reviewed at 48 and 72 h and 5 days after starting the treatment, collecting the report with corresponding antibiogram. Cultivation was the basis for making the decision to change the antibiotic according to the sensitivity and reported resistance. All patients underwent fluid cytology controls.

of PD every 48 hours in hospitalization or by scheduled appointment to PD programs from each hospital. The cytological ones were obtained from a manual exchange (CAPD) with 2 to 4 hours of stay in the cavity without antibiotics to determine the evolution of the symptoms of peritonitis. Through the cytological results and the clinical characteristics, the resolution of the peritonitis. At the beginning and at the end of the peritonitis, biochemical studies were performed: complete blood count (CBC), blood chemistry (QS), serum electrolytes (Na, K, Cl), general urinalysis (EGO) in case of residual urine, culture of site discharge catheter insertion in case of presenting and culture of peritoneal dialysis fluid.

Recorded the clinical features of peritonitis (cloudy PD fluid, abdominal pain, nause).

ELIGIBILITY:
Inclusion Criteria:

* > 18 years in Automated Peritoneal Dialysis.
* Patients in the Hospital General 1, 10 and sub-zone 4 of Colima.
* Patients with diagnosis of peritonitis (abdominal pain, fever, vomiting, nausea, turbid fluid, cytologic with leukocytes >100 cells/mm3, polymorphonuclear >50%).
* Functional catheter.
* Signed informed consent of acceptance to participate in the study.

Exclusion Criteria:

* Patients allergic to vancomicyn.
* Patients allergic to ceftazidime.
* Patients with Intestinal perforation.
* Patients with abdominal cavity classified as unfit to PD.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Trujillo, DS, Study Director — Universidad de Colima
Locations (3):
- Mexico (3):
  - Hgz 10 Instituto Mexicano Del Seguro Social, Manzanillo, Colima
  - Hgsz 4 Instituto Mexicano Del Seguro Social, Tecomán, Colima
  - Hgz 1 Instituto Mexicano Del Seguro Social, Colima

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li PK, Kwong VW. Current Challenges and Opportunities in PD. Semin Nephrol. 2017 Jan;37(1):2-9. doi: 10.1016/j.semnephrol.2016.10.002. PMID 28153192
- [Background] Li PK, Szeto CC, Piraino B, de Arteaga J, Fan S, Figueiredo AE, Fish DN, Goffin E, Kim YL, Salzer W, Struijk DG, Teitelbaum I, Johnson DW. ISPD Peritonitis Recommendations: 2016 Update on Prevention and Treatment. Perit Dial Int. 2016 Sep 10;36(5):481-508. doi: 10.3747/pdi.2016.00078. Epub 2016 Jun 9. No abstract available. PMID 27282851
- [Background] Ruger W, van Ittersum FJ, Comazzetto LF, Hoeks SE, ter Wee PM. Similar peritonitis outcome in CAPD and APD patients with dialysis modality continuation during peritonitis. Perit Dial Int. 2011 Jan-Feb;31(1):39-47. doi: 10.3747/pdi.2009.00235. Epub 2010 Jun 17. PMID 20558813
- [Background] Fielding RE, Clemenger M, Goldberg L, Brown EA. Treatment and outcome of peritonitis in automated peritoneal dialysis, using a once-daily cefazolin-based regimen. Perit Dial Int. 2002 May-Jun;22(3):345-9. PMID 12227392
- [Background] Lan PG, Johnson DW, McDonald SP, Boudville N, Borlace M, Badve SV, Sud K, Clayton PA. The association between peritoneal dialysis modality and peritonitis. Clin J Am Soc Nephrol. 2014 Jun 6;9(6):1091-7. doi: 10.2215/CJN.09730913. Epub 2014 Mar 13. PMID 24626434
- [Background] de Moraes TP, Olandoski M, Caramori JC, Martin LC, Fernandes N, Divino-Filho JC, Pecoits-Filho R, Barretti P. Novel predictors of peritonitis-related outcomes in the BRAZPD cohort. Perit Dial Int. 2014 Mar-Apr;34(2):179-87. doi: 10.3747/pdi.2012.00333. Epub 2014 Jan 2. PMID 24385333
- [Background] El-Reshaid W, Al-Disawy H, Nassef H, Alhelaly U. Comparison of peritonitis rates and patient survival in automated and continuous ambulatory peritoneal dialysis: a 10-year single center experience. Ren Fail. 2016 Sep;38(8):1187-92. doi: 10.1080/0886022X.2016.1209025. Epub 2016 Jul 19. PMID 27435043
- [Background] Sanchez AR, Madonia C, Rascon-Pacheco RA. Improved patient/technique survival and peritonitis rates in patients treated with automated peritoneal dialysis when compared to continuous ambulatory peritoneal dialysis in a Mexican PD center. Kidney Int Suppl. 2008 Apr;(108):S76-80. doi: 10.1038/sj.ki.5002606. PMID 18379553
- [Background] Peerapornratana S, Chariyavilaskul P, Kanjanabuch T, Praditpornsilpa K, Eiam-Ong S, Katavetin P. Short-Dwell Cycling Intraperitoneal Cefazolin Plus Ceftazidime in Peritoneal Dialysis Patients. Perit Dial Int. 2017 Mar-Apr;37(2):218-224. doi: 10.3747/pdi.2015.00300. Epub 2016 Oct 13. PMID 27738089
- [Background] Deslandes G, Gregoire M, Bouquie R, Le Marec A, Allard S, Dailly E, Pineau A, Allain-Launay E, Jolliet P, Roussey G, Navas D. Stability and Compatibility of Antibiotics in Peritoneal Dialysis Solutions Applied to Automated Peritoneal Dialysis in The Pediatric Population. Perit Dial Int. 2016 11-12;36(6):676-679. doi: 10.3747/pdi.2015.00018. Epub 2016 May 4. PMID 27147292
- [Background] Odudu A, Wilkie M. Controversies in the management of infective complications of peritoneal dialysis. Nephron Clin Pract. 2011;118(3):c301-8. doi: 10.1159/000322227. Epub 2011 Jan 14. PMID 21242698
- [Derived] Venegas-Ramirez J, Trujillo-Hernandez B, Castillon-Flores CC, Landin-Herrera FJ, Herrera-Oliva E, Calvo-Soto P, Tapia-Vargas R, Figueroa-Gutierrez A, Rios-Bracamontes EF, Espinoza-Mejia KE, Jimenez-Vieyra IA, Bermudez-Aceves LA, Avila-Flores BJ, Murillo-Zamora E. Simplifying Antibiotic Management of Peritonitis in APD: Evidence from a Non-Inferiority Randomized Trial. Antibiotics (Basel). 2025 Jul 24;14(8):747. doi: 10.3390/antibiotics14080747. PMID 40867942

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 71 patients were diagnosed with peritonitis. 7 patients were excluded because, 5 patients did not meet criteria and 2 voluntary abandonment
Groups:
- Peritonitis Treatment With One Exchange in CAPD: 32 patients in This group will receive peritonitis treatment with one exchange on Continuous Ambulatory Peritoneal Dialysis per day. The initial antibiotic scheme will be with ceftazidime (1500mg/day) and vancomycin (20mg/kg every 3 days) according to current management guidelines; adjusting the management according to the result of the culture, completing the antibiotic scheme for 14 to 21 days.
  Peritonitis treatment with one exchange in CAPD: Antibiotic treatment of peritontiis placed in one bag of Continuos ambulatory peritoneal dialysis per 6 hours each day.
- Peritonitis Treatment Placed in APD: 32 patients in This group will receive peritonitis treatment placed in Automated Peritoneal Dialysis. The initial antibiotic scheme will be with ceftazidime (1500mg/day) and vancomycin (20mg/kg every 3 days); adjusting the management according to the result of the culture, completing the antibiotic scheme for 14 to 21 days.
  Peritonitis treatment placed in APD: Antibiotic treatment of peritontiis placed in bags of Automated peritoneal dialysis.
Period: Overall Study
Arm/Group | Peritonitis Treatment With One Exchange in CAPD | Peritonitis Treatment Placed in APD
Started | 32 | 32
Completed | 32 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Peritonitis Treatment With One Exchange in CAPD: 32 patients in this group will receive peritonitis treatment with one exchange on Continuous Ambulatory Peritoneal Dialysis per day. The antibiotic scheme will be with ceftazidime (1500mg/day) and vancomycin (20mg/kg every 3 days) according to current management guidelines; adjusting the management according to the result of the culture, completing the antibiotic scheme for 14 to 21 days.
  Peritonitis treatment with one exchange in CAPD: Antibiotic treatment of peritontiis placed in one bag of Continuos ambulatory peritoneal dialysis per 6 hours each day.
- Peritonitis Treatment Placed in APD: 32 patiets in this group will receive peritonitis treatment placed in Automated Peritoneal Dialysis, The antibiotic scheme will be with ceftazidime (1500mg/day) and vancomycin (20mg/kg every 3 days); adjusting the management according to the result of the culture, completing the antibiotic scheme for 14 to 21 days.
  Peritonitis treatment placed in APD: Antibiotic treatment of peritontiis placed in bags of Automated peritoneal dialysis.
- Total: Total of all reporting groups
Arm/Group | Peritonitis Treatment With One Exchange in CAPD | Peritonitis Treatment Placed in APD | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Categorical [Count of Participants; unit: Participants] — Population: Lost to follow-up two patients in the intervention group
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 27 | 29 | 56
    >=65 years | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (16.9) | 47.4 (4.6) | 49.42 (72.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 25 | 22 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  spanish race | 32 | 32 | 64
Region of Enrollment [Number; unit: participants]
  Mexico | 32 | 32 | 64
APD modality [Count of Participants; unit: Participants]
  CCPD, continuous cycling peritoneal dialysi | 30 | 29 | 59
  INPD, intermittent nocturnal peritoneal dialysis | 2 | 3 | 5
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.9 (6.0) | 26.6 (4.9) | 27.23 (5.49)
APD per day, duration (hours) [Mean (Standard Deviation); unit: Hours] | 9.6 (0.5) | 9.5 (0.6) | 9.55 (0.56)
Exchanges per day (number) [Mean (Standard Deviation); unit: Exchanges per day (number)] | 5.2 (0.9) | 5.2 (0.8) | 5.2 (0.87)
Tobacco use (yes) [Count of Participants; unit: Participants] | 20 | 18 | 38
Alcohol consumption (yes) [Count of Participants; unit: Participants]
  Alcohol consumption | 24 | 22 | 46
  No Alcohol consumption | 8 | 10 | 18
Type 2 diabetes mellitus (yes) [Count of Participants; unit: Participants] | 21 | 15 | 36
Arterial hypertension (yes) [Count of Participants; unit: Participants] | 31 | 31 | 62
Hypertriglyceridemia (yes [Count of Participants; unit: Participants] | 15 | 19 | 34
Hypercholesterolemia (yes [Count of Participants; unit: Participants] | 16 | 16 | 32
Hyperuricemia (yes) [Count of Participants; unit: Participants] | 8 | 9 | 17
Anemia (yes) [Count of Participants; unit: Participants] | 29 | 29 | 58
Previous peritonitis episode (yes) [Count of Participants; unit: Participants] | 17 | 20 | 37

OUTCOME MEASURES:

1. Primary Outcome: Peritonitis Resolved
Description: We consider the problem resolved when symptoms (nausea, vomiting, abdominal pain, fever, turbid fluid) have disappeared and negative cytology has been obtained (leukocytes <100 cells/mm3)
Time Frame: 14 to 21 days
Population: non-inferiority and the intent-to-treat
Measure: Number; unit: participants
Groups:
- Peritonitis Treatment With ANTIBIOTIC in a Exchange in CAPD + Usual APD: Antibiotic treatment (ceftazidime (1500mg/day) and vancomycin (20mg/kg every 3 days) for 14 to 21 day) into an exchange on CAPD per day + usual APD.
- Peritonitis Treatment Placed in APD: Antibiotic treatment placed in Automated Peritoneal Dialysis bags. (ceftazidime (1500mg/day) and vancomycin (20mg/kg every 3 days) for 14 to 21 days.
Arm/Group | Peritonitis Treatment With ANTIBIOTIC in a Exchange in CAPD + Usual APD | Peritonitis Treatment Placed in APD
Number analyzed (Participants) | 32 | 32
participants | 26 | 29
Statistical Analysis 1: Comparison: Peritonitis Treatment With ANTIBIOTIC in a Exchange in CAPD + Usual APD vs Peritonitis Treatment Placed in APD; Summary statistics were computed, and a significance level (α) of 5% has been established; Test type: Non-Inferiority — The margin of non inferiority analysis was established at 30%; p < 0.05, Chi-squared, Corrected; Risk Ratio (RR) = 1.11, 95% CI 2-sided [0.91 to 1.3], Standard Deviation 95
Statistical Analysis 2: Comparison: Peritonitis Treatment Placed in APD; Test type: Non-Inferiority — margin 30%; p < 0.05, Fisher Exact; Risk Ratio (RR) = 1.0, Standard Deviation 95

2. Secondary Outcome: Death of Patient
Description: Total number and percentage of patients
Time Frame: 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | Peritonitis Treatment With One Exchange in CAPD | Peritonitis Treatment Placed in APD
Number analyzed (Participants) | 32 | 32
Participants | 2 | 2
Statistical Analysis 1: Comparison: Peritonitis Treatment With One Exchange in CAPD vs Peritonitis Treatment Placed in APD; Test type: Non-Inferiority — The margin was established at 30%; p < 0.05, Fisher Exact; Risk Ratio (RR) = 1.0, 1.0% CI 2-sided [0.14 to 6.6], Standard Deviation 95

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Peritonitis Treatment With One Exchange in CAPD | Peritonitis Treatment Placed in APD
All-Cause Mortality (participants affected / at risk) | 2/32 | 2/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT04077996/Prot_SAP_000.pdf